CLINICAL TRIAL: NCT01531803
Title: A Prospective, Randomized, Multicenter, Controlled, Open-Label Study to Evaluate the Safety of Kedbumin25% Compared to Normal Saline Solution in the Treatm. of PostSurgical Hypovolemia in Pediatric Patients Undergoing Major Elective Surgery
Brief Title: Safety Study of Kedbumin 25% Versus Normal Saline in the Treatment of Post-Surgical Hypovolemia in Pediatric Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Per FDA CBER letter dated July 15, 2015, Kedrion SpA was released from the PMC to perform the study with Kedbumin 25% in pediatric patients.
Sponsor: Kedrion S.p.A. (Industry)
Collaborators: inVentiv Health Clinical (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KB058
Record Dates: First submitted 2012-02-01; First posted 2012-02-13 (Estimated); Results first posted 2021-02-18 (Actual); Last update posted 2023-11-15 (Actual); Status verified 2023-10

CONDITIONS: Hypovolemia
MeSH Terms: conditions — Hypovolemia | interventions — Albumins; Saline Solution

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Kedbumin 25% (Experimental): Albumin (Human) 25% solution for intravenous (IV) infusion in the dosage strength of 250g/L human albumin, supplied in 50 mL type II vial (each vial containing 12.5g human albumin).
  The dose will be 0.5 to 1g/kg body weight (2 to 4 mL/kg of 25% albumin). The duration of treatment is based on the subject's response to treatment until hemodynamic stability is achieved. If hemodynamic stability is not achieved within 72 hours of starting the study treatment, the subject will be withdrawn from the study and will be treated according to standard practice and data collected during the study period will be used for the safety evaluation.
  Interventions: Drug: Kedbumin 25%
- Normal Saline Solution (Placebo Comparator): Normal (0.9%) saline solution administered via IV infusions of 10 to 20 mL/kg as appropriate per standard of care based on the subject's clinical status and response to treatment.
  Interventions: Drug: Normal Saline Solution

INTERVENTIONS:
Drug: Kedbumin 25% — Albumin (Human) 25% solution for intravenous (IV) infusion in the dosage strength of 250g human albumin /L, supplied in 50 mL type II vial (each vial containing 12.5g human albumin).
  The dose will be 0.5 to 1g/kg body weight (2 to 4 mL/kg of 25% albumin).
  Other Names: Albumin (Human) 25%
  Arms: Kedbumin 25%
Drug: Normal Saline Solution — Normal (0.9%) saline solution administered via IV infusions of 10 to 20 mL/kg as appropriate per standard of care based on the subject's clinical status and response to treatment.
  Other Names: Normal (0.9%) saline solution
  Arms: Normal Saline Solution

SUMMARY:
This is a randomized, controlled, open-label clinical trial aimed to evaluate the Safety of Kedbumin 25% Compared to Normal Saline Solution in the Treatment of Post-Surgical Hypovolemia in Pediatric Patients Undergoing Major Elective Surgery. It will be conducted at approximately 5 surgical and pediatric intensive care units (SICU/NICU/PICU) in the US, over a period of 19 months, and the study population will consist of at least 60 male and female pediatric subjects between 0 days and 12 years of age, undergoing cardiac, abdominal, orthopedic or transplant surgery with an approximately equal number of subjects (n=10 to 25) in three of the four age groups: (29 days to 23 months), (2 to 5 years 11 months) and (6 years to 12 years) cohorts.

DETAILED DESCRIPTION:
This randomized, controlled, open-label clinical trial will be conducted at approximately 5 surgical and pediatric intensive care units in the US, over a period of 19 months, with 3 months for trial set-up, 12 months of simultaneous subject enrollment and 30 days of treatment/follow-up period, and 3 months for study close-out.

The study population will consist of at least 60 male and female pediatric subjects between 0 days and 12 years of age, undergoing cardiac, abdominal, orthopedic or transplant surgery with an approximately equal number of subjects (n=10 to 25) in three of the four age groups: (29 days to 23 months), (2 to 5 years 11 months) and (6 years to 12 years) cohorts. Regarding the youngest age group of 0 to 28 days, the minimum number of patients to be enrolled in the study will not be predefined as very a small number of elective surgical procedures is expected in this population.

Safety concerns and eventual safety signals, as well as recruitment rate, will be monitored annually (starting from the enrollment of the 60th subject) by an independent Safety Monitoring Board (SMB), which will be appointed prior to study initiation and submitted to the FDA. The responsibilities of the SMB will be defined in ad hoc document, in which the threshold for acceptable safety will also be set. During the conduct of the study on the first 60 patients, if there is any safety signal linked to the primary safety endpoint (i.e. pulmonary fluid overload) or imbalance in the incidence of AEs between the treatment and control groups or based on relevant literature, as judged by the SMB, the enrolment will be increased to 100 patients using the same age stratification approach defined above (n=20 to 30 in each age group).

Potential subjects will be pre-screened and informed consent/assent will be obtained from the subject and/or subject's parents or guardians prior to surgery. Post-surgery, the subject will be admitted to the Surgical, Neonatal, or Pediatric Intensive Care Unit (SICU/NICU/PICU) for post-operative recovery and care management. Subjects who show signs of hypovolemia as judged by the Principal Investigator (PI) will be screened to determine their eligibility to participate in this trial. Subjects will then be randomized to receive treatment with Kedbumin 25% or the comparator, normal saline (sodium chloride 0.9%).

There is no specific post-treatment regimen for this protocol, as all subjects will receive the standard post-operative care based on their clinical status and response to treatment at the discretion of the Investigator.

Vital signs and fluid management/replacement therapy recorded in the medical chart and results of standard complete blood count (CBC), biochemistry, and hematology and coagulation lab panels will be reviewed and recorded by research staff at specified time points, according to the hospital standard of care. Additionally, research staff will review and record daily lactate, urine albumin, blood urea nitrogen (BUN), creatinine, and non-invasive measurements at the following time points: Baseline, 6hr, 12hr, 24hr, 36hr, 48hr, and 72hr post-onset of hypovolemia), until hemodynamic stability is achieved. Hemodynamic stability will be evaluated based on site-specific age-defined reference ranges for heart rate, blood pressure, urine output, and cardiac index in children.

The volume, rate and frequency of the Investigational Medicinal Product (IMP, either Kedbumin 25% or normal saline) administered will be recorded in addition to the type, timing, and amount of all other fluids administered. The time to hemodynamic stability, duration of stability once attained, and any relapse requiring additional treatment or use of secondary resuscitation strategies will be recorded.

Subjects who demonstrate hemodynamic stability within 3 days after treatment initiation and then relapse into hemodynamic instability as a result of surgical complications or infection will exit from the study, but the data be considered for the safety analysis. These subjects should continue treatment according the clinical practice standard since the study is not intended to evaluate the efficacy of Kedbumin 25%.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 0 days to 12 years, inclusive:

   * (0 to 28 days);
   * (29 days to 23 months);
   * (2 to 5 years 11 months);
   * (6 to 12 years).
2. Subjects undergoing elective cardiac, abdominal, orthopedic, or transplant surgery.
3. Subjects with a clinical diagnosis of hypovolemia developed within 24 hours from the completion of surgery, as judged by the Investigator.
4. Admitted to ICU or acute care floor for post-operative recovery and care, in relatively stable condition.
5. Subject, parent or guardian agrees to comply with the requirements of the protocol.
6. Subject, parent or guardian has signed an informed consent form (ICF) and a child assent form if appropriate.
7. Subject, parent or guardian has signed the Health Insurance Portability and Accountability Act (HIPAA) authorization.

Exclusion Criteria:

1. Intra-operative blood loss > 50 mL/kg.
2. Severe hypoalbuminemia with serum albumin levels < 1g/dL.
3. Known intolerance or allergy to albumin and/or plasma proteins.
4. Preterm neonates, defined as neonates with a gestational age of <37 weeks (this criteria would only affect the 0-28 days group).
5. Burn and trauma patients.
6. Renal surgery.
7. Subjects with acute CNS injury or trauma would be excluded from the study.
8. Chronic renal insufficiency or acute renal failure (creatinine > 1.5 of normal value or based on age-appropriate renal function parameters), or a history of renal transplantation.
9. Subjects with hypernatremia, defined as a Na level of ≥ 155 mEq/L.
10. Severe congestive heart failure (CHF) using one of the following classification systems: Ross Heart Failure Classification, modified Ross Heart Failure Classification, or New York University Pediatric Heart Failure Index (NYU PHFI).
11. Any concurrent medical, surgical or psychiatric condition that may, in the Investigator's opinion, affect the subject's ability to meet the protocol requirements.
12. Subject has participated in another interventional clinical study within 30 days prior to study enrollment. Subjects who are participating in another observational study are not excluded.

Max Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2015-02-05 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2015-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mirella Calcinai, MD, Study Director — Kedrion SpA
Locations (2):
- United States (2):
  - Kosair Charities Pediatric Unit, Louisville, Kentucky
  - Medical College of Wisconsin, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Kedbumin 25%: Albumin (Human) 25% solution for intravenous (IV) infusion in the dosage strength of 250g/L human albumin, supplied in 50 mL type II vial (each vial containing 12.5g human albumin).
  The dose will be 0.5 to 1g/kg body weight (2 to 4 mL/kg of 25% albumin). The duration of treatment is based on the subject's response to treatment until hemodynamic stability is achieved. If hemodynamic stability is not achieved within 72 hours of starting the study treatment, the subject will be withdrawn from the study and will be treated according to standard practice and data collected during the study period will be used for the safety evaluation.
  Kedbumin 25%: Albumin (Human) 25% solution for intravenous (IV) infusion in the dosage strength of 250g human albumin /L, supplied in 50 mL type II vial (each vial containing 12.5g human albumin).
  The dose will be 0.5 to 1g/kg body weight (2 to 4 mL/kg of 25% albumin).
Period: Overall Study
Arm/Group | Kedbumin 25% | Normal Saline Solution
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This study has been prematurely stopped. Only 3 participants have been enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Kedbumin 25% | Normal Saline Solution | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 2 | 3
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence, Severity, and Seriousness of Fluid Overload and Edema (Pulmonary Portal or Systemic) and/or Other Complications Secondary to Fluid Resuscitation With Kedbumin 25% Compared to Normal Saline.
Description: Criteria for Primary Evaluation:
  1. Presence of rales at pulmonary bases: cut-off YES/NO and at least one of the following:
     * Chest X Ray: presence of Kerley B lines: cut-off YES/NO;
     * Doppler sonography to measure the pulmonary artery pressure: cut-off >20mmHg;
     * Arterial oxygen saturation: cut-off ≤ 90% and/or ABG: cut-off pO2 ≤ 70mmHg.
  2. Fluid overload and edema is quantified by % increase in body weight over the subject's preoperative weight stratified by <10%, 11-15%, 16-20% and >20%.
  3. Physical examination for edema.
  All the measurements for the assessment of the safety parameters will be collected, reviewed, and recorded by research staff until hemodynamic stability is achieved.
Time Frame: 3 days
Population: The study has been prematurely stopped.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedbumin 25% | Normal Saline Solution
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

2. Secondary Outcome: Resolution of Hypovolemia With Adequate Fluid Resuscitation and Restoration of Hemodynamic Stability After Treatment With Kedbumin 25% Compared to Normal Saline Within 72 Hours.
Description: The secondary safety parameter of resolution of hypovolemia and adequate fluid resuscitation will be evaluated based on the following indicators:
  * Hemodynamic status [heart rate (HR), blood pressure (BP), urine output (UOP)];
  * Tissue hypoperfusion [lactate levels, base deficit derived from arterial blood gas, if arterial line is in place] or determined by the use of a pulse oximetry;
  * Electrolyte status [Na+, Ca++, Mg++, K+, Cl- ,PO4];
  * Renal/hepatic function [urine albumin, blood urea nitrogen (BUN), creatinine, creatinine clearance, total bilirubin, ALT, AST, Albumin, Alkaline Phosphatase (ALP), gamma glutamyltransferase (GGT)];
  * Complete blood count (CBC);
  * Partial Thromboplastin Time/ International Normalized Ratio (PTT/INR).
  All the measurements for the assessment of the safety parameters will be collected, reviewed, and recorded by research staff until hemodynamic stability is achieved.
Time Frame: 3 days
Population: The study has been prematurely stopped.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedbumin 25% | Normal Saline Solution
Number analyzed (Participants) | 1 | 2
Participants | 0 | 0

3. Secondary Outcome: Incidence, Severity and Seriousness of Expected and Unexpected AEs After Treatment With Kedbumin 25% Compared to Normal Saline.
Description: The severity, seriousness, and relatedness of AEs to the study drug will be observed on repeated administrations of the study drug.
  Subjects will be carefully monitored by the SICU/NICU/PICU or acute care floor staff for expected and unexpected AEs which occur from the time of dosing to 30 days post dose.
  If the subject is discharged prior to 30 days, research staff will collect AEs at follow-up visits and via spontaneous reporting by the subject.
Time Frame: 30 days
Population: The study has been prematurely stopped. Only 3 participants have been enrolled and one of them showed a non-serious adverse event (AE) of superficial wound infection of mild intensity not related to the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Kedbumin 25% | Normal Saline Solution
Number analyzed (Participants) | 1 | 2
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Arm/Group | Kedbumin 25% | Normal Saline Solution
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Kedbumin 25% (N=1) | Normal Saline Solution (N=2)
Superficial Wound Infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Superficial wound infection of mild intensity. The subject was treated with 22.68 mg clindamycin intravenous every 6 hours (18 Feb 2015 to 23 Feb 2015). The AE resolved on 23 Feb 2015 and was considered to be not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No